CLINICAL TRIAL: NCT01145014
Title: A Randomised, Double-blind, Placebo-controlled (Within Dose Groups) Phase I - Study to a) Assess Safety, Tolerability and Pharmacokinetics of Single Rising Oral Doses 2 mg to 600 mg of BI 660848 Administered as Oral Drinking Solution (Powder in Bottle) in Healthy Male Volunteers, b) to Explore the Relative Oral Bioavailability of an Immediate Release Tablet Formulation and c) to Assess the Impact of a High Fat Meal on the Oral Bioavailability of the Oral Drinking Solution (Powder in Bottle).
Brief Title: To Investigate Safety, Tolerability, and Pharmacokinetics of Treatment With BI 660848 Rising Single Doses (From 2 mg to 600 mg) Administered as Oral Drinking Solution (Powder in Bottle).
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Boehringer Ingelheim, Study Chair, Boehringer Ingelheim
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1284.1; 2009-015995-90 (EudraCT Number: EudraCT)
Record Dates: First submitted 2010-05-05; First posted 2010-06-16 (Estimated); Last update posted 2013-11-01 (Estimated); Status verified 2013-10

CONDITIONS: Pain; Healthy
MeSH Terms: conditions — Pain

ARMS (12):
- BI 660848 2 mg (Experimental): oral drinking solution
  Interventions: Drug: BI 660848
- BI 660848 10 mg (Experimental): oral drinking solution
  Interventions: Drug: BI 660848
- BI 660848 20 mg (Experimental): oral drinking solution
  Interventions: Drug: BI 660848
- BI 660848 50 mg (Experimental): oral drinking solution
  Interventions: Drug: BI 660848
- BI 660848 100 mg (Experimental): oral drinking solution
  Interventions: Drug: BI 660848
- BI 660848 150 mg (Experimental): oral drinking solution
  Interventions: Drug: BI 660848
- BI 660848 200 mg (Experimental): oral drinking solution
  Interventions: Drug: BI 660848
- BI 660848 400 mg (Experimental): oral drinking solution
  Interventions: Drug: BI 660848
- BI 660848 600 mg (Experimental): oral drinking solution
  Interventions: Drug: BI 660848
- BI 660848 10,0 mg (Experimental): immediate release tablet
  Interventions: Drug: BI 660848
- BI 660848 50,0 mg (Experimental): immediate release tablet
  Interventions: Drug: BI 660848
- Placebo (Experimental): matching placebo (oral drinking solution and IR tablets)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: BI 660848 — 2 mg oral drinking solution
  Arms: BI 660848 2 mg
Drug: BI 660848 — 10 mg oral drinking solution
  Arms: BI 660848 10 mg
Drug: BI 660848 — 20 mg oral drinking solution
  Arms: BI 660848 20 mg
Drug: BI 660848 — 50 mg oral drinking solution
  Arms: BI 660848 50 mg
Drug: BI 660848 — 100 mg oral drinking solution
  Arms: BI 660848 100 mg
Drug: BI 660848 — 150 mg oral drinking solution
  Arms: BI 660848 150 mg
Drug: BI 660848 — 200 mg oral drinking solution
  Arms: BI 660848 200 mg
Drug: BI 660848 — 400 mg oral drinking solution
  Arms: BI 660848 400 mg
Drug: BI 660848 — 600 mg oral drinking solution
  Arms: BI 660848 600 mg
Drug: BI 660848 — 10,0 mg immediate release tablet
  Arms: BI 660848 10,0 mg
Drug: BI 660848 — 50,0 mg immediate release tablet
  Arms: BI 660848 50,0 mg
Drug: Placebo — matching placebo (oral drinking solution and IR tablets)
  Arms: Placebo

SUMMARY:
As a transition from preclinical investigations to clinical development in this first-in-human trial, safety, tolerability, and pharmacokinetics of BI 660848 will be assessed in human male volunteers using single rising oral doses in order to provide the basis for a potential ongoing clinical development of BI 660848 in the indication of neuropathic pain.

ELIGIBILITY:
Inclusion criteria

1. Healthy male based upon a complete medical history, including the physical examination, regarding vital signs (BP, PR), 12 lead ECG measurement, and clinical laboratory tests. There is no finding deviating from normal and of clinical relevance. There is no evidence of a clinically relevant concomitant disease.
2. Age 21 and 50 years
3. BMI 18.5 and <30 kg/m2 (Body Mass Index)
4. Signed and dated written informed consent prior to admission to the study in accordance with GCP and the local legislation

Exclusion criteria

1. Any finding of the medical examination (including BP, PR, and ECG measurements) deviating from normal and of clinical relevance
2. Evidence of a clinically relevant concomitant disease
3. Gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders
4. Diseases of the central nervous system (such as epilepsy) or psychiatric disorders or neurological disorders
5. History of relevant orthostatic hypotension, fainting spells or blackouts
6. Chronic or relevant acute infections
7. History of relevant allergy/hypersensitivity (including allergy to the drug or its excipients) as judged clinically relevant by the investigator
8. Intake of drugs with a long half-life (24 hours) within at least 1 month or less than 10 half-lives of the respective drug prior to randomisation
9. Use of drugs which might reasonably influence the results of the trial based on the knowledge at the time of protocol preparation within 10 days prior to randomisation
10. Participation in another trial with an investigational drug within 2 months prior to randomisation
11. Smoker (>10 cigarettes or >3 cigars or >3 pipes/day)
12. Inability to refrain from smoking on trial days as judged by the investigator
13. Alcohol abuse (more than 30 g alcohol a day)
14. Drug abuse
15. Blood donation (more than 100 mL blood within 4 weeks prior to randomisation or during the trial)
16. Excessive physical activities within 1 week prior to randomisation or during the trial
17. Any laboratory value outside the reference range that is of clinical relevance
18. Inability to comply with dietary regimen of the study centre

Ages: 21 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 72 (Actual)
Dates: Start 2010-05; Primary Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability (number and intensity of adverse events). | 4 months
Changes in blood pressure. | 4 months
Changes in pulse rate. | 4 months
Changes in respiratory rate. | 4 months
Changes in 12-lead ECG. | 4 months
Changes in clinical laboratory test parameters. | 4 months

SECONDARY OUTCOMES:
Cmax (maximum measured concentration of the analyte in plasma) | 3 days
tmax (time from dosing to maximum measured concentration) | 3 days
AUC (area under the concentration-time curve of the analyte in plasma over the time interval from 0 extrapolated to infinity) | 3 days
t1/2 (terminal half-life of the analyte in plasma) | 3 days
MRT (mean residence time of the analyte in the body after drug intake) | 3 days
CL/F (apparent clearance of the analyte in plasma after extravascular administration) | 3 days
Vz/F (apparent volume of distribution during the terminal phase following an extravascular dose) | 3 days
Aet1-t2 (amount of analyte eliminated in urine from the time point t1 to time point t2) | 3 days
fet1-t2 (fraction of analyte eliminated in urine from the time point t1 to time point t2) | 3 days
CL R,t1-t2 (renal clearance of the analyte from the time point t1 until the time point t2) | 3 days

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (1):
- 1284.1.1 Boehringer Ingelheim Investigational Site, Ingelheim, Germany